CLINICAL TRIAL: NCT00245973
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of Bifeprunox in the Treatment of Depression in Outpatients With Bipolar Disorder
Brief Title: Study Evaluating Bifeprunox in Bipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3168A2-307
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Depression Bipolar
MeSH Terms: conditions — Bipolar Disorder | interventions — bifeprunox

INTERVENTIONS:
Drug: Bifeprunox

SUMMARY:
The purpose of the study is to investigate whether eight weeks of treatment with flexible doses of Bifeprunox is superior to treatment with placebo in depressed patients with bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 65 years of age, inclusive.
* Diagnosis of Bipolar Disorder and must be experiencing a depressive episode.

Exclusion Criteria:

* This is a follow on study to protocol 3168A2-304. Only subjects who have participated in the previous study are eligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380
Dates: Start 2005-06; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Secondary measurement scales will be used:
Hamilton Psychiatric Rating Scale for Depression (HAM-D17), at baseline, and weeks 1, 2, 3, 4, 6, and 8

SECONDARY OUTCOMES:
Clinical Global Impressions Severity of Illness Score (CGI-S),at screening, baseline, and weeks 1, 2, 3, 4, 6, and 8
Clinical Global Impressions Improvement Score (CG-I), at weeks 1, 2, 3, 4, 6, and 8
Young-Mania Rating Scale (Y-MRS), at screening, baseline, and weeks 1, 2, 3, 4, 6, and 8
Positive and Negative Symptom Scale (PANSS) at at screening, baseline, and weeks 1, 2, 3, 4, 6, and 8
Covi Anxiety Scale at screening, baseline, and weeks 2, 4, 6, and 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (39):
- United States (39):
  - Birmingham, Alabama
  - Beverly Hills, California
  - National City, California
  - Stanford, California
  - Farmington Hills, Connecticut
  - Bradenton, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - West Palm Beach, Florida
  - Smyrna, Georgia
  - Honolulu, Hawaii
  - Terre Haute, Indiana
  - Florence, Kentucky
  - New Orleans, Louisiana
  - Rockville, Maryland
  - Boston, Massachusetts
  - Farmington Hills, Michigan
  - Saint Charles, Missouri
  - Clementon, New Jersey
  - Moorestown, New Jersey
  - Lawrence, New York
  - New York, New York
  - Staten Island, New York
  - The Bronx, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Lyndhurst, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Salt Lake City, Utah
  - Bellevue, Washington
  - Seattle, Washington
  - Brown Deer, Wisconsin